CLINICAL TRIAL: NCT00311337
Title: Evaluation of Safety and Efficacy of VELCADE as Maintenance Treatment in Patients With Multiple Myeloma Following High-Dose Melphalan Treatment and Autologous PBSCT (Minimal Residual Disease, Partial Remission or Stable Disease)
Brief Title: VELCADE as Maintenance Treatment in Patients With Multiple Myeloma Following Autologous Peripheral Blood Stem Cell Transplantation (PBSCT)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuerzburg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSMM VIII
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2006-04-05 (Estimated); Status verified 2006-03

CONDITIONS: Multiple Myeloma
Keywords: VELCADE; bortezomib; maintenance treatment; multiple myeloma; primary disease
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
Protocol DSMM VIII is a multi-center, open-label study evaluating the safety and tolerability, as well as the efficacy, of maintenance treatment with VELCADE (bortezomib) in patients with multiple myeloma with detectable disease activity following tandem high-dose chemotherapy and autologous SCT. The time from SCT to the initiation of VELCADE treatment will be 3 to 6 months.

DETAILED DESCRIPTION:
Protocol DSMM VIII is a multi-center, open-label study evaluating the safety and tolerability, as well as the efficacy, of maintenance treatment with VELCADE in patients with multiple myeloma with detectable disease activity following tandem high-dose chemotherapy and autologous SCT. The time from SCT to the initiation of VELCADE treatment will be 3 to 6 months.

The initial 11 patients entered into this trial will be treated at a dose level of 1.0 mg/m2 once weekly on 4 consecutive weeks followed by 2 weeks of rest. A total of 4 treatment cycles is planned.

An interim analysis for safety and tolerability will be performed after at least the first cycle of study drug has been completed. If the study treatment is found to be safe and no dose-limiting toxicity has occurred, the dose of VELCADE will be increased to 1.3 mg/m2 and another 11 patients will be treated at this dose level according to the treatment schedule as outlined above. The dose escalation to 1.3 mg/m2 will be performed without delay if no AE or SAE are reported to the principal investigator.

If the safety of a specific dose level is acceptable the efficacy of the maintenance treatment will be statistically evaluated. The treatment is considered to be efficacious if a minimum of 25% of all treated patients experience a success, considered as remission of their disease within 6 months after the end of VELCADE treatment. The therapy will be acceptable for further clinical studies if a minium of 25% successfully treated patients will be observed.

Under these assumptions in the first step of the optimal two step design (Simon 1989) 21 patients have to be treated. As patients included during phase I are included in the efficacy analysis, this means an additional 10 patients to be treated. If less than three patients were successfully treated defined as an improvement in the remission status, the study will be stopped, because the success rate is unacceptably low. If three or more of the 21 patients are successfully treated, another 29 patients will be included. At the end of the study the success rate will be evaluated. If 8 or more of the 50 patients were successfully treated the therapy will be acceptable for further studies.

Patients will be evaluated at scheduled screening and baseline visits. After providing written informed consent to participate in the study, patients will be screened for study eligibility during a screening period of 28 days. Baseline assessment consists of a detailed history of pre-existing diseases, blood tests including disease-specific markers such as ß2-microglobulin, IgG, IgA, IgM, immunofixation from blood and urine, serum free light chains, a bone marrow biopsy, a skeletal survey, an electrocardiogram and a chest X-ray.

The study drug will be administered in study centers only. Prior to each administration of study drug, a short medical history focusing on VELCADE-associated side effects will be performed as well as complete blood cell counts, kidney and liver function tests.

A visit on day 30 following the last administration of study drug for the final assessment of safety and tolerability is mandatory in all patients included in this protocol.

Serological myeloma specific markers (monoclonal immunoglobulin, serum free light chains and immunofixation from blood and urine) will be performed at weeks 6, 12, 18 and 24 and thereafter in 3 months intervals. Bone marrow biopsies will be performed when serological markers indicate complete remission or progression, a skeletal survey once a year during follow-up. During the study, disease will be assessed according to the EBMT/IBMTR/ABMTR criteria.

Safety will be evaluated by the occurrence of clinical and laboratory toxicities and changes from baseline in physical examination findings, vital signs, and, if applicable, chest X-ray and electrocardiogram findings. All patients will receive an aminobisphosphonate at 4 weekly intervals. Other disease-modifying treatment such as alpha interferon or pulsed corticosteroids are strictly prohibited.

ELIGIBILITY:
Inclusion Criteria:

* Patient having received tandem transplants with high-dose melphalan and autologous PBSCT within 3-6 months prior to inclusion into this protocol
* Patients with measurable minimal residual disease (very good partial remission [VGPR]) or patients in partial remission (PR) or patients with stable disease (SD) at the time of inclusion in the study
* Patient must agree to participate in the study.
* Patient agrees to use an appropriate method of contraception.
* Willingness and ability to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Patient showing signs of disease progression
* Patient has a platelet count < 100 x 10^9/L within 14 days before enrollment.
* Patient has an absolute neutrophil count < 1.0 x 10^9/L within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance < 30 mL/minute within 14 days before enrollment.
* Patient has >= Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has hypersensitivity to bortezomib, boron, or mannitol.
* Patient has received prior treatment with bortezomib
* Patient is pregnant or nursing
* Patient has received other investigational drugs within 14 days before enrollment
* Patient has progressive disease
* Patient has a Karnofsky performance status < 60%
* Patient has a life expectancy of < 3 months
* Patient has received disease modifying agents following autologous stem cell transplantation other than aminobisphosphonates such as interferon-alpha or glucocorticosteroids
* Patient currently enrolled in another clinical research study and/or receiving an investigational reagent for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61
Dates: Start 2005-10; Study Completion 2010-10

PRIMARY OUTCOMES:
Primary endpoints are to study the safety of four cycles of VELCADE in patients with multiple myeloma following high-dose chemotherapy and autologous PBSCT.

SECONDARY OUTCOMES:
The secondary objectives of this study are to assess the efficacy of four cycles of VELCADE at two different dose levels as maintenance treatment in patients with multiple myeloma
and detectable residual disease following high-dose chemotherapy and autologous PBSCT
to assess the 2 year progression-free survival
and to assess the 2 year overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Einsele, MD, Principal Investigator — Dept. of Internal Medicine II, University of Wuerzburg, Klinikstr. 6-8, 97070 Wuerzburg; Hermann Einsele, MD, Principal Investigator — Dept. of Internal Medicine, University of Wuerzburg
Locations (8):
- Austria (2):
  - Medizinische Univ.-Klinik Graz, Graz
  - Klin. Abt. für Onkologie, AKH Wien, Vienna
- Germany (5):
  - Dept. of Hematology/Oncology, Charité Berlin, Berlin
  - Dept. of Internal Medicine, Ludwig-Maximilian-University Munich, Munich
  - Dept. of Internal Medicine A, University Muenster, Münster
  - Dept. of Internal Medicine III, University of Ulm, Ulm
  - Dept. of Internal Medicine II, University of Wuerzburg, Würzburg
- Regionalkrankenhaus Bozen, Bolzano, Italy